CLINICAL TRIAL: NCT00570271
Title: Physiological Effects of Placebo Interventions to Increase or Decrease Blood Pressure
Brief Title: Placebo Effects on Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Dr. H.-C. Deter, Dept of Psychosomatic Medicine and Psychotherapy, Benjamin Franklin Campus, Charité,Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EA4/004/07; EA4/004/07
Record Dates: First submitted 2007-12-05; First posted 2007-12-10 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-11

CONDITIONS: Blood Pressure
Keywords: placebo effect; blood pressure; autonomic nervous system; prestige; basic research on physiological placebo effects
MeSH Terms: interventions — Desoxycorticosterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental)
  Interventions: Other: Placebo with BP dec (written form)
- 2 (Experimental)
  Interventions: Other: Placebo with BP dec (doctor)
- 3 (Experimental)
  Interventions: Other: Placebo with BP inc (written)
- 4 (Experimental)
  Interventions: Other: Placebo with BP inc (doctor)
- 5 (No Intervention)
  Interventions: Other: Placebo info given (written)
- 6 (No Intervention)
  Interventions: Other: Placebo info given (doc)

INTERVENTIONS:
Other: Placebo with BP dec (written form) — Placebo administration with a blood pressure decrease suggestion. Information provided to subjects in written form.
  Arms: 1
Other: Placebo with BP dec (doctor) — Placebo administration with a blood pressure decrease suggestion. Information provided to subjects by doctor.
  Arms: 2
Other: Placebo with BP inc (written) — Placebo administration with a blood pressure increase suggestion. Information provided to subjects in written form.
  Arms: 3
Other: Placebo with BP inc (doctor) — Placebo administration with a blood pressure increase suggestion. Information provided to subjects by doctor.
  Arms: 4
Other: Placebo info given (written) — Subject informed about receiving placebo. Information provided to subjects in written form.
  Arms: 5
Other: Placebo info given (doc) — Subject informed about receiving placebo. Information provided to subjects by doctor.
  Arms: 6

SUMMARY:
A relevant reduction of blood pressure (BP) in placebo-treated control groups is a phenomenon often observed in pharmacological studies of hypertension. This effect was shown to differ from spontaneous remission tendencies and regression to the mean effect by comparing placebo groups with untreated controls. However, it is not fully understood whether these effects are due to a global reaction of the autonomous nervous system (affecting the overall organ systems of the body) or a specific reaction (affecting the cardiovascular system only). We therefore aim to differentiate specific effects (reduction of blood pressure) from global effects (e.g. changes in electrodermal and gastric activity).

In our study we aim to test the following hypotheses:

1. Placebo administration leads to a significant changes of blood pressure compared with untreated controls.
2. The direction of blood pressure change depends on the type of suggestion (either decrease or increase)
3. This effect is specific for blood pressure; changes in electrodermal and gastric activity do not differ between groups.
4. The placebo response can be enhanced by a prestige intervention (information about the suggested drug action given by doctor or in written form).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent

Exclusion Criteria:

* Not meeting inclusion criteria
* Untreated hypertension (BP > 140/90) or hypotension(BP < 100/60)
* Severe systemic disorders (tumors, tbc, diabetes, asthma etc)
* Diseases with influence on cardiovascular or gastrointestinal system
* Pregnancy and lactation phase
* Body mass index > 30
* Regular intake of drugs with influence on the autonomic nervous system
* Insufficient compliance
* Simultaneous participation in another trial

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-04; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure | 60 minutes

SECONDARY OUTCOMES:
Heart rate | 60 minutes
skin conductance level | 60 minutes
gastric activity | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christian Deter, MD, Study Director — Charité University Berlin
Locations (1):
- Department of Psychosomatic Medicine and Psychotherapy, Charité University, Berlin, Germany